CLINICAL TRIAL: NCT01932814
Title: Retrospective Analysis of Aminoglycoside-associated Acute Renal Injury in Septic Critically Ill Patients
Brief Title: Acute Kidney Injury in Septic Critically Ill Patients : Are Aminoglycosides Really Harmful?
Acronym: REAMICHOC
Status: Completed | Type: Observational
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Responsible Party: Principal Investigator, Alexandre Boyer, MD,phD, Université Victor Segalen Bordeaux 2
Other Study IDs: REAMICHOC
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Acute Kidney Injury; Severe Sepsis
Keywords: Aminoglycosides; Acute kidney injury; Severe sepsis; Critically ill patient
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aminoglycosides: have received aminoglycosides
- No Aminoglycosides: did not receive aminoglycosides

SUMMARY:
The purpose of the present study is to determine whether administration of aminoglycosides in septic critically ill patient is a risk factor for acute kidney injury

DETAILED DESCRIPTION:
Severe sepsis and septic shock despite recent advances in surviving sepsis campaign remain encumbered by a high mortality rate close to 30%. One cornerstone of the management of these patients remains the early and appropriate antibiotic administration, , which must be also active at the site of infection. Aminoglycosides are often administered in combination with beta lactams in this context . According to the progress in pharmacokinetic management achieved over the past decade, their safety and efficiency tended to increase but many uncertainties remain. The purpose of the present study is to determine whether administration of aminoglycosides in septic critically ill patient is a risk factor for acute kidney injury.

Study design: This is an open retrospective monocentric cohort study including septic critically ill patients from november 2008 to january 2010. To determine the incidence and the specific risk of nephrotoxicity of aminoglycosides, only hospitalized patients without initial acute kidney injury or with rapidly improving kidney function during the three first days will be included.Primary outcome will be the occurrence of acute kidney injury assessed with the RIFLE classification (Risk, Injury, Failure, Loss, and End-stage kidney disease) from day 4 to day 15. Patients receiving aminoglycosides will be compared with a control group, i.e. not receiving them. We estimated hazard ratios (HR) and 95% confidence intervals (CI) with adjusted and propensity score (PS)-matched Cox-proportional hazards models.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Admission to ICU with severe sepsis
* Hospitalized and without acute kidney injury or with kidney function improved on the third day were included
* Information provided to the patient or proxy

Exclusion Criteria:

* Renal replacement therapy before day 3
* Patients with renal insufficiency J1 (Day 1 creatinine clearance <56.25 ml/mn/1, 73m2) but severely altered between Day 1 and Day 3 (creatinine clearance Day 1/ Day 3> 1 + Day 3 creatinine clearance <37.5 ml/mn/1, 73m2 ) without renal replacement therapy still necessary before J3
* Prolonged aminoglycosides therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill septic patients
Sampling Method: Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The incidence of acute renal injury associated with treatment with aminoglycoside in critically ill septic patients | between day 4 and day 15

SECONDARY OUTCOMES:
Risk factors of acute kidney injury | between day 1and day 3

OTHER OUTCOMES:
Risk factors for ICU mortality | between day 4 and day 15
Pharmacokinetics parameters of aminoglycosides | between day 1 to day 6
  daily dose, peak serum concentration, through level serum concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation médicale, Hôpital Pellegrin, Bordeaux, Aquitaine, France

REFERENCES:
- [Result] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Result] Boucher BA, Coffey BC, Kuhl DA, Tolley EA, Fabian TC. Algorithm for assessing renal dysfunction risk in critically ill trauma patients receiving aminoglycosides. Am J Surg. 1990 Nov;160(5):473-80. doi: 10.1016/s0002-9610(05)81007-4. PMID 2240380
- [Result] Boyer A, Gruson D, Bouchet S, Clouzeau B, Hoang-Nam B, Vargas F, Gilles H, Molimard M, Rogues AM, Moore N. Aminoglycosides in septic shock: an overview, with specific consideration given to their nephrotoxic risk. Drug Saf. 2013 Apr;36(4):217-30. doi: 10.1007/s40264-013-0031-0. PMID 23508544
- [Result] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Result] Kollef MH, Sherman G, Ward S, Fraser VJ. Inadequate antimicrobial treatment of infections: a risk factor for hospital mortality among critically ill patients. Chest. 1999 Feb;115(2):462-74. doi: 10.1378/chest.115.2.462. PMID 10027448
- [Result] Kumar A, Safdar N, Kethireddy S, Chateau D. A survival benefit of combination antibiotic therapy for serious infections associated with sepsis and septic shock is contingent only on the risk of death: a meta-analytic/meta-regression study. Crit Care Med. 2010 Aug;38(8):1651-64. doi: 10.1097/CCM.0b013e3181e96b91. PMID 20562695